CLINICAL TRIAL: NCT05570708
Title: The Role of Personal Experience for the Therapeutic Attitude in the Context of Substance-assisted Therapy Training
Acronym: TherPsySE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Felix Mueller (Other)
Collaborators: Swiss Medical Society for Psycholytic Therapy (Other)
Responsible Party: Sponsor-Investigator, Felix Mueller, Sponsor-Investigator PD Dr. med. Felix Müller MD, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-01173
Record Dates: First submitted 2022-09-21; First posted 2022-10-07 (Actual); Last update posted 2025-04-14 (Actual); Status verified 2025-04

CONDITIONS: Personal Experience of Substance-assisted Therapy Using Psilocybin, MDMA, and LSD
MeSH Terms: interventions — N-Methyl-3,4-methylenedioxyamphetamine; Lysergic Acid Diethylamide; Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personal experience of substance-assisted therapy using psilocybin, MDMA, and LSD (Experimental)
  Interventions: Drug: MDMA, LSD, psilocybin

INTERVENTIONS:
Drug: MDMA, LSD, psilocybin — * MDMA per os (2 x 100mg) in a group setting
  * LSD per os (75 and 150 mcg) in a 1:1 setting
  * Psilocybin per os (15 mg and 25 mg) in a group setting
  * Three study days are without drug administration: Participants experience the role of the therapist in a 1:1 setting

SUMMARY:
The study investigates two groups of participants of the SÄPT therapist's training starting in October 2022. The overall objective is to investigate the risks and benefits of personal experience (PE) with substance-induced altered states of consciousness for physicians or psychotherapists in the context of a training course for substance-assisted therapy. Specifically, the study aims to assess changes in therapeutic attitude and other factors important in interactions between patients and therapists (such as empathy and cognitive flexibility).

ELIGIBILITY:
Inclusion Criteria:

* Participation in the SÄPT therapist training (medical doctors and psychologists)
* Age 27 years or older
* Sufficient understanding of the German language
* Understanding of procedures and risks associated with the study
* Willing to adhere to the protocol and signing of the consent form
* Willing not to operate heavy machinery (including driving cars) within 24 hours after substance administration
* Woman of childbearing potential are required to use effective, established contraception, such as oral, injected or implanted hormonal methods of contraception, placement of an intrauterine device (IUD) or intrauterine system (IUS), barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository at least one month before and after each study substance intervention, and are willing to take a urine pregnancy test at the medical screening and before every study substance intervention.
* Men are required to use contraceptive methods in the month after each study substance intervention and are required to inform their partner(s) about their study participation.

Exclusion Criteria:

* Previous significant adverse response to a hallucinogenic drug
* Significant medical condition rendering volunteers unsuitable for participation (such as impaired kidney or liver function, or heart disease incl. uncontrolled hypertension or hypotension)
* Strong underweight (<45kg)
* Current major psychiatric disorder (including personality disorder, including suicidality) and / or previous psychotic or bipolar disorder.
* Psychotic disorder or bipolar disorder in first-degree relatives
* Use of medication that may interfere with the effects of the study medication. Patients must be willing to discontinue medications in cases where drug-related interactions are possible (the washout phase will be at least 5 times the particular drug's half-life [typically 3-7 days] prior to the respective study session). Discontinuation of medication must be judged to be acceptable by the responsible investigator.
* Women are excluded from substance intervention during pregnancy or breastfeeding.
* nParticipation in another clinical trial (currently or within the last 30 days)

Min Age: 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
TASC-2 scale | Three weeks after last PE
  The primary endpoint is changes on the TASC-2 scale of the Therapeutic attitude questionnaire (ThAT)

SECONDARY OUTCOMES:
semi-structured interview | Five months after last PE
  A semi-structured interview will be used to explore the range of effects and systematically collect and record subjective effects of the personal experience
TASC-2 scale | Three weeks after each PE and six months after last PE
  TASC-2 scale of the Therapeutic attitude questionnaire (ThAT)
SOCS-S | Three weeks after each PE and six months after last PE
  Compassion with self
SPCS-O | Three weeks after each PE and six months after last PE
  Compassion with others
SPF/IRI | Three weeks after each PE and six months after last PE
  Empathy questionnaire
5D-ASC | Directly after each PE
  5 dimensions of altered states of consciousness questionnaire
CEQ | Directly after each PE
  Challenging experience questionnaire
APEQ | Directly after each PE
  Acceptance /avoidance-promoting experiences questionnaire
PIQ | Directly after each PE
  Psychological insights questionnaire
CSOWD | Directly after each PE
  Connectedness scale
EBI | Directly after each PE
  Emotional breakthrough inventory
BFW/E | Three weeks after each PE and six months after last PE
  Berner Subjective Well-Being questionnaire
PEQ | Three weeks after each PE and six months after last PE
  Persisting effects questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Felix Müller, MD, Principal Investigator — University of Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No